CLINICAL TRIAL: NCT00670696
Title: A Randomised, Controlled, Single-blinded, Cross Over Comparison Study to Compare the Efficacy of the Rapydan Medicated Plaster Versus Tetracaine Gel
Brief Title: A Study to Compare the Efficacy of Rapydan Versus Tetracaine Gel
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No longer sponsor of trial
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RD 305/24674
Record Dates: First submitted 2008-04-29; First posted 2008-05-02 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Healthy; Anesthesia
Keywords: Topical anesthesia; Rapydan; Topical anaesthesia for venous cannulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Rapydan medicated plaster administered 30 minutes prior to cannulation on Visit 1 and tetracaine gel administered 45 minutes prior to cannulation on Visit 2.
  Interventions: Drug: Rapydan
- B (Active Comparator): Tetracaine gel administered 45 prior to cannulation on Visit 1 and then Rapydan administered 30 minutes prior to cannulation on Visit 1
  Interventions: Drug: tetracaine gel

INTERVENTIONS:
Drug: Rapydan — Topical anaesthetic plaster
  Arms: A
Drug: tetracaine gel — Topical tetracaine gel
  Arms: B

SUMMARY:
Tetracaine gel 4% is a topical anaesthetic gel commonly used in the UK that contains 40 mg of tetracaine base per gram. Adequate anaesthesia can usually be achieved following a 30 minute application time for venopuncture and a 45 minute application time for venous cannulation. The hypothesis is that Rapydan medicated plaster is more effective than tetracaine gel in preventing venous cannulation related pain when applied for the recommended treatment durations of 30 minutes and 45 minutes respectively.

DETAILED DESCRIPTION:
Tetracaine gel 4% is a topical anaesthetic gel commonly used in the UK that contains 40 mg of tetracaine base per gram. Adequate anaesthesia can usually be achieved following a 30 minute application time for venopuncture and a 45 minute application time for venous cannulation. The hypothesis is that Rapydan medicated plaster is more effective than tetracaine gel in preventing venous cannulation related pain when applied for the recommended treatment durations of 30 minutes and 45 minutes respectively. This study has been withdrawn and no additional data is available.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects of any race, 18 yrs or older
* No clinically significant findings on physical exam
* Signed informed consent

Exclusion Criteria:

* Damaged, denuded or broken skin at the designated site for application of the medicated plaster or gel.
* Know allergies to lidocaine, tetracaine or other local anaesthetics
* Concomitant use of prescription strength analgesics

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-04; Primary Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
To demonstrate superiority for Rapydan medicated plaster applied 30 minutes over tetracaine gel applied for 45 minutes in terms of reducing pain associated with venous cannulation as assessed by the subject on a 100 mm visual analog scale (VAS) | VAS post venous cannulation

SECONDARY OUTCOMES:
To demonstrate comparable tolerability between Rapydan medicated plaster and tetracaine gel | Up to 14 days post exposure

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Dimber, MD, Principal Investigator — EUSA Pharma, Inc.
Locations (1):
- Merthyr Tydfill Industrial Estate, Merthyr, Tydfill, United Kingdom